CLINICAL TRIAL: NCT01990391
Title: Effect of Brazil Nut Consumption in the Microvascular Endothelial Function, Oxidative Stress and Metabolic Abnormalities in Hypertensive and Dyslipidemic Subjects
Brief Title: Brazil Nut Consumption in Microvascular Endothelial Function, Oxidative Stress and Metabolic Abnormalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Instituto Nacional de Cardiologia de Laranjeiras (Other); Oswaldo Cruz Foundation (Other); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Grazielle Vilas Boas Huguenin, Mrs, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0008.0.197.185-11; U1111-1132-2061 (Other: Universal trial number)
Record Dates: First submitted 2013-11-10; First posted 2013-11-21 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Dyslipidemia; Oxidative Stress
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cassava flavored flour (Placebo Comparator): The placebo group (cassava flour flavored) received 9g/day of cassava flour flavored during three months (12 weeks)
  Interventions: Dietary Supplement: Brazil nut flour
- Brazil nut flour (Experimental): The Brazil nut group received 13g/day of Brazil nut flour during three months (12 weeks)
  Interventions: Dietary Supplement: Placebo (cassava flavored flour)

INTERVENTIONS:
Dietary Supplement: Brazil nut flour — The Brazil nut group received 13g/day of Brazil nut flour during three months.
  Arms: Cassava flavored flour
Dietary Supplement: Placebo (cassava flavored flour) — The group placebo (cassava flour flavored)received 9g/day of cassava flour flavored during three months
  Arms: Brazil nut flour

SUMMARY:
The purpose this research is to check the effect of Brazil Nuts consumption in oxidative stress, metabolic abnormalities and microvascular endothelial function dyslipidemic and hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* adults > 20 years old
* Dyslipidemic
* Hypertensive

Exclusion Criteria:

* Allergy to nuts
* Consumption of nuts or vitamins/minerals supplement
* Loss weight before the research
* pregnancy
* Kidney chronic disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Antioxidant biomarker | Change from Baseline at 12 weeks.
  Change from Baseline plasma Gluthathione Peroxidase activity (nmol/min/ml) at 12 weeks, samples were stocked at -80 degrees.

SECONDARY OUTCOMES:
Oxidative stress biomarker | Change from Baseline at 12 weeks.
  The change from baseline plasma 8-isoprostane (pg/ml) at 12 weeks, samples were stocked at -80 degrees.
microvascular endothelial function | Change from baseline at 12 weeks
  Microvascular reactivity was evaluated using an Laser Speckle Contrast Imaging system with a laser wavelength of 785 nm in combination with the iontophoresis (increasing anodal currents of 30, 60, 90, 120, 150 and 180μA for 10 second intervals spaced 1 minute apart) of acetylcholine (2% v/v) for the noninvasive and continuous measurement of cutaneous microvascular perfusion changes measured in arbitrary perfusion units.

OTHER OUTCOMES:
Anthropometric measures | Change from baseline at 12 weeks
  body weight (kg), body mass index (kg/m2) and waist circumference (cm).
Blood lipids | Change from baseline at 12 weeks
  total Cholesterol (mg/dl), LDL-cholesterol (mg/dl), HDL-cholesterol (mg/dl) and triglycerides (mg/dl).

CONTACTS AND LOCATIONS:
Overall Officials: Grazielle V B Huguenin, Nutricionist, Principal Investigator — Universidade Federal do Rio de Janeiro

REFERENCES:
- [Derived] Carvalho RF, Huguenin GV, Luiz RR, Moreira AS, Oliveira GM, Rosa G. Intake of partially defatted Brazil nut flour reduces serum cholesterol in hypercholesterolemic patients--a randomized controlled trial. Nutr J. 2015 Jun 16;14:59. doi: 10.1186/s12937-015-0036-x. PMID 26077768
- [Derived] Huguenin GV, Oliveira GM, Moreira AS, Saint'Pierre TD, Goncalves RA, Pinheiro-Mulder AR, Teodoro AJ, Luiz RR, Rosa G. Improvement of antioxidant status after Brazil nut intake in hypertensive and dyslipidemic subjects. Nutr J. 2015 May 29;14:54. doi: 10.1186/s12937-015-0043-y. PMID 26022214